CLINICAL TRIAL: NCT03909555
Title: Effects of Short-term Intensive Insulin Therapy on Long-term Complications in Patients With Type 2 Diabetes
Brief Title: Effects of Short-term Intensive Insulin Therapy on Long-term Complications in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Zhujiang Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Jinan University (Other); Guangzhou Red Cross Hospital (Other); Dongguan Kanghua Hospital (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology and Metabolism Department, Sun Yat-sen University
Other Study IDs: 20181015
Record Dates: First submitted 2019-01-21; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Continuous subcutaneous insulin infusion; chronic complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short-term intensive insulin therapy: Patients who used to participated in short-term intensive insulin therapy for 14 days when diabetes was newly diagnosed
  Interventions: Other: Complications assessment
- Routine diabetic therapy: Received routine diabetic therapy
  Interventions: Other: Complications assessment

INTERVENTIONS:
Other: Complications assessment — Records of cardiovascular diseases (CVD), carotid ultrasonography, electrocardiogram, echocardiography, fundus photography, urinary albumin excretion, Toronto Clinical Neuropathy Scale and Composite Autonomic Symptom Score.

SUMMARY:
Short-term intensive insulin therapy (SIIT) is able to reverse β cell dysfunction and induce glycemic remission in patients with newly diagnosed type 2 diabetes. On the other hand, intensive control of glucose and lifestyle modification are two key elements in preventing chronic complications, especially microvascular neuropathy. However, no study reported the long-term effect of SIIT on the chronic complications. In this multi-center, case-control study, effects of SIIT on the proportion of long-term chronic complications as well as potential biomarkers were investigated.

In total, 777 patients with type 2 diabetes, including 259 patients who participated SIIT when diabetes was newly diagnosed and 518 patients who received routine diabetic therapy will be enrolled in 12 centers in China. After baseline assessments, all patients will undergo complications assessment, including records of cardiovascular diseases (CVD), carotid ultrasonography, electrocardiogram, echocardiography, fundus photography, urinary albumin excretion, Toronto Clinical Neuropathy Scale and Composite Autonomic Symptom Score. Primary endpoint is the difference in the proportions of macrovascular and microvascular complications between groups. Secondary endpoints include the difference of glucose control, insulin resistance, complexity of anti-diabetic therapy and self-management skills and quality of life between two groups. What's more, new biomarkers, which may indicate the occurrence of chronic complications of diabetes, such as circulating endothelial progenitor, β cell dysfunction, and T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as type 2 diabetes for at least 5 years;
2. When diagnosed as diabetes for the first time, aged between 25 and 65 years, body mass index (BMI) 22-35 kg/m2, fasting plasma glucose (FPG) between 7.0 mmol/l (126 mg/dl) and 16.7 mmol/l (300 mg/dl);
3. Short-term intensive insulin therapy group: Patients received short-term intensive insulin therapy for 14 days when newly diagnosed as type 2 diabetes and induce glycemic remission.
4. Routine diabetic therapy group: Patients received routine diabetic therapy as guideline indicated and never induce glycemic remission.

Exclusion Criteria:

1. Type 1 diabetes or special type of diabetes;
2. Acute complications of diabetes (including DKA, HHS and lactic acidosis) when diagnosed as diabetes;
3. Serious microvascular complications: proliferative stage of retinopathy; urine AER >300 mg/g or urine protein positive, quantification >0.5 g/d; uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy when diagnosed as diabetes;
4. Severe macrovascular complications: acute cerebrovascular accident, acute coronary syndrome, vascular intervention for peripheral arterial disease or amputation requiring hospitalization within 12 months prior to enrollment when diagnosed as diabetes;
5. Blood creatinine clearance less than 50 ml/min, alanine aminotransferase ≥2.5×upper limit of normal, total bilirubin ≥1.5×upper limit of normal; Hemoglobin <100 g/L or need regular blood transfusion;
6. Use of drugs that may influence blood glucose within 12 weeks;
7. Systemic infection or serious concomitant disease; patients with malignancy or chronic diarrhea;
8. Uncontrolled endocrine gland dysfunction;
9. Patients with mental or communication disorders;
10. Chronic cardiac insufficiency, heart function class III and above;
11. Pregnant women, lactating women and women of child bearing age who are not willing to take contraception during the study;
12. Subjects who don't cooperate, cannot be followed up or have difficulty in completing the study considered by the investigator.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 777 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportions of chronic complications | 5 year
  Difference in the proportions of macrovascular and microvascular complications between groups

SECONDARY OUTCOMES:
Difference of glycosylated hemoglobin A1C | 5 year
  Difference of glycosylated hemoglobin A1C between groups
Difference of fast blood glucose | 5 year
  Difference of fast blood glucose between groups
Difference of C-peptides | 5 year
  Difference of fast C-peptides between groups.
Difference of insulin resistance | 5 year
  Difference of HOMA2-IR between groups. HOMA2-IR is calculated by fast blood glucose and C-peptide according to formula proposed by DR Matthew (the software can be accessed at http://www.ocdem.ox.ac.uk).
Difference of insulin usage | 5 year
  Compare the proportion of insulin usage (including rapidly acting insulin, regular insulin, long-acting insulin and premixed insulin) between groups
Difference of oral anti-diabetic drugs usage | 5 year
  Compare the proportion of oral anti-diabetic drugs usage (including biguanides, sulfonylureas, Glinides, glucosidase inhibitors, thiazolidinediones, DPP 4 inhibitors, SGLT-2 inhibitor and their combination) between groups
Difference of attitudes toward diabetes | 5 year
  Compare the score of Diabetes Care Profile questionnaire between groups. Patients were questioned about five aspects, including positive attitude, negative attitude, ability to care for their diabetes, belief in importance of care, and self-care adherence. Each statement included a 5-point ranking scale, ranging from strongly disagree (never) to strongly agree (always), with 3 points as neutral. Items under the subscales of positive attitude, care ability, importance of care, and self-care adherence scoring ≥4 points and items of negative attitude scoring≤2 points were designated as good performance, whereas the opposites were poor.
Difference of quality of life | 5 year
  Compare the score of Diabetes quality of life (DQOL) between groups. The DQOL contains a total of 46 items, and all the items are categorized into one of the following four domains: life satisfaction (15 items), diabetes impact (20 items), social/vocational related worries (7 items), and diabetes related worries (4 items). The DQOL adopts a 5-point Likert scale for its response options. The scores range from 1, labeled as "very satisfied," to 5, labeled as "very dissatisfied," for items in the life satisfaction domain; from 1, labeled as "never impacted," to 5, labeled as "always impacted," for items in the diabetes impact domain; and from 1, labeled as "never worried," to 5, labeled as "always worried," for the social/vocational related and diabetes related worries domains. Higher score indicating better outcome.

OTHER OUTCOMES:
New biomarkers which may indicate the occurrence of chronic complications of diabetes | 5 year
  Proportion of circulating endothelial progenitor cells between groups. Low level of circulating endothelial progenitor cells indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided